CLINICAL TRIAL: NCT06237361
Title: Muscle Strength, Functional Capacity and Quality of Life Responses to Pilates Exercises in Children With Burn Injuries
Brief Title: Pilates Benefits in Pediatric Burn Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Collaborators: Prince Sattam Bin Abdulaziz University (Other); Cairo University (Other)
Responsible Party: Principal Investigator, Maged Basha, Associate Professor, College of Medical Rehabilitation, Qassim University, Qassim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/023/014
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Burns; Pilates Exercise; Pediatric Burn
MeSH Terms: conditions — Burns | interventions — Exercise Movement Techniques; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional physical therapy programs (Experimental): group that received traditional physical therapy programs (TPTP) alone
  Interventions: Other: traditional physical therapy program
- Pilates group (Experimental): received both traditional physical therapy programs and Pilates exercises.
  Interventions: Other: Pilates exercises; Other: traditional physical therapy program

INTERVENTIONS:
Other: Pilates exercises — participants underwent a 12-week intervention involving three Pilates sessions per week. The Pilates exercises comprised warm-up activities, Pilates routines, and cool-down exercises.
  Other Names: Pilates band
  Arms: Pilates group
Other: traditional physical therapy program — The program included a variety of exercises such as range of motion exercises, aerobic exercises, resistance exercises, scar management, occupational therapy, and hand therapy.
  Other Names: Exercise

SUMMARY:
This study investigated the effects of Pilates exercises on lower limb muscle strength, functional capacity, and quality of life in children with burn injuries. In a twelve-week randomized clinical trial involving 60 children, those who received Pilates exercises in addition to traditional physical therapy showed significant improvements in muscle strength, functional capacity, and overall quality of life compared to those who received traditional therapy alone. The findings suggest that incorporating Pilates exercises into rehabilitation programs may enhance outcomes for children recovering from burn injuries.

DETAILED DESCRIPTION:
This research focused on examining the impact of Pilates exercises on lower limb muscle strength, functional capacity, and quality of life in children recuperating from burn injuries. The study, conducted as a twelve-week randomized clinical trial with 60 participants, found notable improvements in various aspects for the group receiving Pilates exercises alongside traditional physical therapy. Specifically, enhancements in muscle strength (including hip flexors, extensors, abductors, and more), functional capacity, and overall quality of life scores were statistically significant in the Pilates group compared to those undergoing traditional therapy alone. This suggests a positive influence of Pilates exercises on the rehabilitation of children with lower limb burns.

The investigation delved into the potential benefits of Pilates exercises, emphasizing their role in augmenting muscle strength, functional capacity, and overall well-being. The study participants, aged 10 to 15 years and recovering from lower limb burns, were randomly assigned to either a control group receiving only traditional physical therapy or a Pilates group combining Pilates exercises with traditional therapy. The outcomes demonstrated significant differences favoring the Pilates group, not only in terms of lower limb muscle strength but also functional capacity, as assessed by the 6-minute walk test, and overall quality of life scores measured through the Pediatric Quality of Life Inventory. The findings suggest that incorporating Pilates into rehabilitation programs for pediatric burn survivors can contribute positively to physical and functional recovery, potentially improving their overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

Children with lower limb (LL) healed burns. Age between 10 and 15 years. Six months post-injury. Mixed deep 2nd & 3rd degree burn. Total body surface area (TBSA) between 35-55 percent. Capability to walk securely without assistance.

Exclusion Criteria:

Lower limb joint range of motion limits. Mental illnesses. Significant behavioral or cognitive impairments. Incapacity to exercise. Metabolic diseases. Neuropathy. Visual or vestibular abnormalities. Medical instability.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-10-22 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Muscle Strength Assessment | at baseline
  Assessed using a calibrated handheld dynamometer (Micro FET2, Hoggan Health Technologies Inc., UT, USA), participants performed three 5-second contractions for each muscle group. The average score in newtons was calculated for each muscle group.
Muscle Strength Assessment | after 12 weeks
  Assessed using a calibrated handheld dynamometer (Micro FET2, Hoggan Health Technologies Inc., UT, USA), participants performed three 5-second contractions for each muscle group. The average score in newtons was calculated for each muscle group.
6-minute walk test | at baseline
  Participants were timed and given six minutes to walk as far as they could along a straight course. Running, jumping, or hopping were not allowed.
6-minute walk test | after 12 weeks
  Participants were timed and given six minutes to walk as far as they could along a straight course. Running, jumping, or hopping were not allowed.

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory | at baseline
  A self-report questionnaire assessing the health-related quality of life (HRQL) of children and adolescents. It includes physical health, psychosocial health, and a total summary score.
Pediatric Quality of Life Inventory | after 12 weeks
  A self-report questionnaire assessing the health-related quality of life (HRQL) of children and adolescents. It includes physical health, psychosocial health, and a total summary score.

CONTACTS AND LOCATIONS:
Overall Officials: Alshimaa Azab, PhD, Study Chair — Professor, Faculty of Physical Therapy, Cairo University; Maged Basha, PhD, Study Director — Qassim University
Locations (1):
- Outpatient Clinic of College of Applied Medical Sciences, Prince Sattam bin Abdulaziz University, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Background] Aibar-Almazan A, Martinez-Amat A, Cruz-Diaz D, Jesus de la Torre-Cruz M, Jimenez-Garcia JD, Zagalaz-Anula N, Redecillas-Peiro MT, Mendoza-Ladron de Guevara N, Hita-Contreras F. The Influence of Pilates Exercises on Body Composition, Muscle Strength, and Gait Speed in Community-Dwelling Older Women: A Randomized Controlled Trial. J Strength Cond Res. 2022 Aug 1;36(8):2298-2305. doi: 10.1519/JSC.0000000000003790. Epub 2020 Sep 25. PMID 32991508
- [Result] Farrell RT, Gamelli RL, Sinacore J. Analysis of functional outcomes in patients discharged from an acute burn center. J Burn Care Res. 2006 Mar-Apr;27(2):189-94. doi: 10.1097/01.BCR.0000202615.59734.0E. PMID 16566563
- [Result] Gojowy D, Kauke M, Ohmann T, Homann HH, Mannil L. Early and late-recorded predictors of health-related quality of life of burn patients on long-term follow-up. Burns. 2019 Sep;45(6):1300-1310. doi: 10.1016/j.burns.2019.03.016. Epub 2019 Jun 5. PMID 31176508
- [Derived] Azab AR, Basalem N, Alghadier M, Khanam H, George J, Aloraini SM, Alsultan F, Basha MA, S Waked I, Kamel FH. Muscle Strength, Functional Capacity, and Quality of Life Responses to Pilates Exercises in Children with Burn Injuries: A Single-Blinded Randomized Clinical Trial. Iran J Med Sci. 2025 Nov 1;50(11):743-753. doi: 10.30476/ijms.2025.104947.3852. eCollection 2025 Nov. PMID 41262321